CLINICAL TRIAL: NCT07072702
Title: Feasibility and Acceptability of an Evidence-Informed Virtual Intervention to Reduce Perceptions of Injustice Following Work Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Michael Sullivan, Principal investigator, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SULL2024
Record Dates: First submitted 2025-05-08; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: MSK Conditions
Keywords: Pain; Disability; Psychosocial; Perceived Injustice
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This feasibility study will use a 4-centre (clinic), single arm, prospective design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MPIC (Experimental): A brief evidence-informed intervention was developed to reduce post-injury perceptions of injustice. The intervention is referred to as 'Managing Post-Injury Challenges' (MPIC). MPIC consists of 4 weekly 30-minute virtual meetings with a psychologist trained in the delivery of the intervention. MPIC is delivered concurrently with the physiotherapy treatment to which the injured worker has been referred. MPIC combines elements of validation, motivational interviewing, acceptance and problem-solving.
  Interventions: Behavioral: Managing Post-Injury Challenges (MPIC)

INTERVENTIONS:
Behavioral: Managing Post-Injury Challenges (MPIC) — A brief evidence-informed intervention was developed to reduce post-injury perceptions of injustice. The intervention is referred to as 'Mastering Post-Injury Challenges' (MPIC). MPIC consists of 4 weekly 30-minute virtual meetings with a psychologist trained in the delivery of the intervention. MPIC is delivered concurrently with the physiotherapy treatment to which the injured worker has been referred. MPIC combines elements of validation, motivational interviewing, acceptance and problem-solving .

SUMMARY:
Many individuals who have sustained disabling injuries in the workplace react to their situation with a sense of 'injustice'. Research over the past 20 years has revealed that, interpreting one's post-injury life situation as 'unjust', actually interferes with recovery from the disabling injury. Post-injury perceptions of injustice contribute to more severe pain, more severe symptoms of depression and PTSD, and more prolonged absence from work. Several clinical researchers have highlighted the need to develop approaches to treatment that can reduce post-injury perceptions of injustice.

A brief intervention was developed to reduce post-injury perceptions of injustice. The intervention consists of 4 30-minute sessions with a psychologist. The intervention is called 'Managing Post-Injury Challenges' (MPIC). The MPIC sessions are delivered virtually (online). As a first step toward determining whether MPIC has added value for promoting more successful recovery following work injury, the proposed research will assess the feasibility of MPIC. Some of the feasibility questions that will be addressed include: Are injured workers interested in participating in MPIC? Do injured individuals remain sufficiently engaged to complete all 4 sessions of MPIC? Does participation in MPIC contribute to meaningful reductions in perceived injustice? And are injured individuals satisfied with the benefits of MPIC?

MPIC differs from many other rehabilitation interventions in that it focuses on a 'risk-factor' for problematic recovery as opposed to treating a specific health or mental health problem. At this time, there is little information about whether injured workers are interested in interventions focusing on 'risk factors' for problematic recovery. As a first step in evaluating the effectiveness of MPIC, it is necessary to demonstrate that MPIC is acceptable to injured workers. We would consider the study to be successful if 1) at least 75% of eligible injured workers agree to enrol in MPIC, 2) if at least 75% of participants attend all 4 sessions of MPIC, and if at least 75% of participants are satisfied with the benefits they derived from their involvement in MPIC. If MPIC is ultimately shown to be effective in reducing post-injury perceptions of injustice, offering MPIC to injured workers with elevated scores on a measure of perceived injustice could contribute to more successful recovery.

DETAILED DESCRIPTION:
There is increasing evidence that perceptions of injustice can contribute to adverse recovery outcomes in individuals with disabling musculoskeletal conditions. Individuals who obtain elevated scores on measures of perceived injustice also report more severe pain, reduced participation in important activities of daily living, prolonged work disability, and the persistence of symptoms of mental health problems such as depression and post-traumatic stress disorder. Recent reviews of the literature have concluded that perceptions of injustice are strong predictors of disability and depression in individuals with musculoskeletal conditions. The emerging pattern of findings suggests that perceived injustice triggers a cascade of cognitive (i.e., rumination), emotional (anger, depression) and behavioural (i.e., activity withdrawal, medication overuse) reactions that can impede recovery. The relation between perceived injustice and adverse recovery outcomes has been demonstrated in individuals with work-related low back pain, whiplash injuries, catastrophic injuries, traumatic head injuries, fibromyalgia, sickle cell disease , osteoarthritis, and rheumatoid arthritis.

Although there are currently no intervention programs that have been developed specifically to modify perceptions of injustice following work injury, there are indications that treatment-related reductions in perceptions of injustice are prospectively associated with more positive rehabilitation outcomes. For example, one study reported that reductions in perceptions of injustice predicted occupational re-engagement in work-disabled individuals participating in a 10-week behavioural activation program. In the latter study, reductions in perceived injustice predicted return to work even when controlling for treatment-related reductions in pain severity. In a separate study, treatment-related reductions in perceptions of injustice were found to prospectively predict reductions in depressive symptom severity in work-disabled individuals with Major Depressive Disorder. The research that has accumulated to date suggests that an intervention specifically designed to reduce perceptions of injustice could contribute to more positive recovery outcomes in individuals who have sustained debilitating musculoskeletal injuries.

The purpose of the proposed study is to test the feasibility and impact of a 4-week psychosocial intervention, delivered remotely, designed to reduce perceptions of injustice following occupational injury. The intervention consists of 4 30-minute virtual meetings with a psychologist trained in the delivery of the intervention protocol. The intervention protocol has been termed, 'Managing Post-Injury Challenges' (MPIC). The intervention protocol is manualized and combines several evidence-supported treatment elements including validation, motivational interviewing, acceptance and problem-solving. The intervention protocol will be delivered concurrently with physiotherapy treatment.

Participants

The study sample will consist of 75 individuals who are absent from work due to a musculoskeletal injury. All participants will be receiving primary care physical therapy from one of 4 clinics. Eligibility criteria will include 1) receiving or having applied for time-loss benefits from the WSIB for a musculoskeletal injury to the back or neck, 2) date of injury less than 6 weeks prior to enrolment in the study, 3) a score above risk threshold on a self-report measure of perceived injustice, and 4) working knowledge of French or English. Individuals who are currently receiving psychological treatment will not be considered for participation.

Measures

All self-report measures will be administered through a secure web-based data capture system (RedCap).

Demographic and Injury-Related Variables. Participants will be asked to complete a general information form where they will be asked to respond to questions concerning their age, sex, education, marital status, number of children at home, occupation, previous time loss claims and current medication intake.

Perceived injustice: The Injustice Experiences Questionnaire (IEQ) will be used to measure injury-related perceptions of injustice.

Pain Severity: The McGill Pain Questionnaire Short-Form (MPQ-SF) will be used to measure pain severity.

Depressive symptoms: The Patient Health Questionnaire-9 (PHQ-9) will be used to assess depressive symptom severity. Self-Reported Disability: The WHODAS 2.0 will be used to assess self-rated disability.

Treatment satisfaction will be assessed at treatment termination. Return to Work. Return-to-work status will be assessed by telephone interview at treatment termination and 3-month follow-up.

Procedure

Consecutive referrals meeting the inclusion criteria for the study will be invited to participate. Prospective participants will be provided with a brief description of the intent of the MPIC intervention and will be asked for permission to be contacted by one of the MPIC clinicians. Prospective participants who agree to participate in the MPIC intervention will be provided with a link to a secure portal that will be used to administer all self-report measures used in the proposed research. MPIC sessions will be scheduled at a mutually convenient time for the MPIC clinician and the participants, and will be held weekly for 4 consecutive weeks. All self-report measures will be administered at the time of enrollment in the study (Week 1), at termination of the MPIC intervention (Week 4) and at 3-month follow-up. Treatment satisfaction will only be assessed at termination of the MPIC intervention.

A post-treatment debriefing interview will be conducted at 3-month follow-up. The aim of the post-treatment interview will be to examine participants' reflections on aspects of the intervention that they considered beneficial and aspects of the intervention that they did not consider beneficial. These interviews will provide important information to guide possible modifications to the intervention protocol that could increase its engagement value and impact.

The short-term expected outcome is that we will demonstrate that MPIC will yield clinically significant reductions in perceived injustice. We also expect that the results of the study will show that reductions in perceived injustice predict more positive recovery outcomes.

The next step in the evolution of this program of research would be to confirm the effectiveness of MPIC within the context of a randomized controlled trial. The long-term expected outcome is that there will be interest from the clinical practice community to acquire the skill set required to deliver the MPIC intervention.

The telehealth model of service delivery also has several advantages over face-to-face treatment including ease of incorporation into other health services to which participants might have been referred, physical accessibility, geographical reach, low cost, and feasibility of quality monitoring. The advantages of combining a risk-targeted intervention with an accessible service delivery model, while minimizing displacement challenges for individuals with a disabling health condition might provide the optimal approach for reducing the pain, disability and chronicity that can ensue in the aftermath of work injury.

It is anticipated that the study findings will reveal that the risk-targeted intervention yields meaning reductions in perceived injustice, and in turn, contributes to more positive recovery outcomes. Such findings would support the addition of the risk-targeted intervention to the repertoire of services made available to injured workers. The telehealth delivery model would maximize the scalable potential of the intervention to meet the needs of the target population. Training modules could be developed to disseminate the skill set required to deliver the intervention to the broader clinical practice community.

ELIGIBILITY:
Inclusion Criteria:

1. working knowledge of English,
2. work absence of less than 8 weeks duration following a musculoskeletal injury to the back or neck,
3. a score above clinical threshold on a self-report measure of perceived injustice,
4. between 25 and 65 years of age,
5. referred for primary care physiotherapy, and
6. currently receiving wage indemnity benefits from the WSIB.

Exclusion Criteria:

1. currently receiving psychological services for a mental health problem,
2. clinical evidence of vertebral fracture, disk herniation, infectious disease, or rheumatoid arthritis (determined from referral information),
3. illiteracy or severe cognitive impairment (determined informally through the intake interview).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceived Injustice | The IEQ will be administered pre-treatment, treatment termination and 3-month follow-up.
  The Injustice Experiences Questionnaire (IEQ) will be used to assess post-injury perceptions of injutice.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request.